CLINICAL TRIAL: NCT02802800
Title: A Comparison of Land Based and Water Based Plyometric Training Effects on the Physical Fitness of Field Hockey Players in Jamaica
Brief Title: A Comparison of Land and Water Based Plyometric Training on Fitness of Field Hockey Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Sharmella Roopchand-Martin, Lecturer, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECP214-13-14
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Fitness Training
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water (Experimental): Plyometric Training in water, twice per week for 6 weeks.
  Interventions: Other: Plyometric training
- Land (Experimental): Plyometric training on land, twice per week for 6 weeks.
  Interventions: Other: Plyometric training

INTERVENTIONS:
Other: Plyometric training — Plyometric exercises
  Other Names: Power training

SUMMARY:
Field hockey players, recruited from clubs in Jamaica, will be randomized to either a water training or land training groups. Persons will be exposed to 6 weeks of plyometric training with two sessions per week. Pre and post test measures will be done for lower limb power, flexibility and agility. Distance covered, pace, heart rates and exertion during a match will also be assessed.

DETAILED DESCRIPTION:
Plyometric training has been used in a variety of sports to improve power. There is minimal research however regarding its use among hockey players and even less research exploring water based training. International field hockey competitions are played on wet turf and it is felt that water training may be beneficial to these players. The study will explore whether water based plyometrics will prove to have additional benefits compared to land based plyometrics for the Jamaican hockey athletes. The members of the Jamaica hockey clubs will be recruited to participate in this study. Recruitment will be done by the principal investigator Dr. Roopchand-Martin. A total of 34 persons will be recruited and they will be randomly allocated to aquatic or land based training. All training programmes will be conducted at the section of physical therapy and training will be done two times per week for 6 weeks. Baseline assessments will be done independent evaluators for lower limb power using the Standing Broad Jump and Vertical Jump Test, anaerobic power using the Running Anaerobic Sprint test, agility using the Illinois agility and T tests, flexibility using the Sit and Reach Test and performance during game play on wet artificial turf in relation to time-motion analysis for total distance covered, and total time, average and maximum pace, average and maximum heart rate, time in heart zones 1-5, and changes in rate of perceived exertion.

ELIGIBILITY:
Inclusion Criteria:

* All club hockey players over the age of 16 in Kingston and St. Andrew, Jamaica

Exclusion Criteria:

* Persons with musculoskeletal injuries of the hip or knee, who have undergone surgery or injections in the past 3 months, or who are under rehabilitation and not at the phase to undergo high intensity training will be excluded.
* Persons with skin diseases, open wounds and self-reported aqua phobia will also be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 6 weeks
  Vertical jump will be measured using the Brower vertical jump apparatus. The standing height with one arm extended upward is recorded and then the athlete jumps off two feet and the sensor on the bar records the jump height. Each person will complete 3 jumps and the best trial recorded. The jump height recorded is the difference between the jump height and the standing reach height.
Standing Broad Jump | 6 weeks
  Participant will stand with feet together and then jump forward as far as they can. The trials will be completed and the best jump recorded. Distance jumped will be measured with a tape measure.
Illinois Agility Test scores | 6 weeks
  Participants will be asked to run through a course marked out on the hockey field. The best of two trials will be recorded. Timing of the trials will be done using the Brower TC timing gate system.
Agility T test | 6 weeks
  Participants will complete a course that is marked out on the hockey field. Two trials will be done and the best trial time recorded. Timing will be done with a stopwatch
Sit and Reach Distance | 6 weeks
  Participants with sit on a bed with legs outstretched and their back and buttock against a wall. They will place one hand over the other and then be asked to reach forward as far as they can without bending their knees. Three trials will be allowed and the furthers reach distance recorded.

SECONDARY OUTCOMES:
Distance covered during a match | 6 weeks
  Distance run during a a match will be captured with the Polar M400 sports watch GPS trackers which participants will wear during 30 minutes of competition.
Heart rate during a match | 6 weeks
  Heart rate during a 30 minute match will be captured with the Polar M400 sports watch with GPS trackers and heart rate monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Therapy, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: No